CLINICAL TRIAL: NCT03754712
Title: Effect of Vitamin D Administration Along With Selective Serotonin Reuptake Inhibitors (SSRIs) in Patients With Major Depressive Disorder (MDD)
Brief Title: Effect of Vitamin D Administration Along With SSRIs in Patients With Major Depressive Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh (Other)
Responsible Party: Principal Investigator, Tanzina Afrin, MD, Resident, Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: No. BSMMU /2018/2964
Record Dates: First submitted 2018-11-25; First posted 2018-11-27 (Actual); Last update posted 2018-11-28 (Actual); Status verified 2018-11

CONDITIONS: MDD
MeSH Terms: interventions — Cholecalciferol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Vitamin D3 along with SSRIs (Active Comparator): One tablet of vitamin D3 (2000IU) per day for 8 weeks
  Interventions: Dietary Supplement: Vitamin D3
- SSRIs (No Intervention): Patients treated with SSRIs

INTERVENTIONS:
Dietary Supplement: Vitamin D3 — Dietary supplement : Vitamin D3 one tablet of vitamin D3 (2000IU) per day for 8 weeks
  Arms: Intervention Vitamin D3 along with SSRIs

SUMMARY:
Several studies suggested low serum levels of vitamin D have been associated with depression. So, the present study is designed to investigate the effect of vitamin D administration along with SSRIs in patients with MDD.

DETAILED DESCRIPTION:
Depression is a major global health problem. Major depression was ranked as the third leading cause of the global burden of diseases in 2004 and is supposed to occupy the first place by 2030. Major depression is a complex and multifactorial symptom-complex while dysfunctions in various endocrine axes may be independent risk factors in the development of the affective illness. Some recent observations indicate a significant role of vitamin D regarding mood. Vitamin D3 receptors have been found in cerebral cortex, cerebellum, and the limbic system. The active form of vitamin D on the nervous system is associated with modifying the production and release of neurotrophic factors such as nerve growth factor (NGF) which is essential for neuron differentiation, as well as increasing the levels of glial cell line derived neurotrophic factor (GDNF). Vitamin D influence the expression of genes associated GABA-ergic neurotransmission. It also stimulates the expression of tyrosine hydroxylase which is responsible for catecholamines biosynthesis. Lately, positive influences of vitamin D upon patients suffering from MDD have been suggested. This area require further attention and confirmation as little work has been carried out in this field. So, the present study is an attempt to investigate the effect of vitamin D administration along with SSRIs in patients with MDD. The study would be a interventional one to be conducted in the department of Pharmacology and in the department of psychiatry, BSMMU. A total of 90 patients suffering from major depression will be selected according to inclusion and exclusion criteria. The diagnosis of patients suffering from major depression and the selection of SSRIs would be performed by medical officer of the Psychiatry department. After completing necessary formalities including informed consent of the patients, patient's data will be collected to measure baseline complaints of depression. The patients would be divided into two groups: group A and B. Group A would consist of 45 patients who will receive only SSRIs and Group B would consist of 45 patients who will receive SSRIs plus vitamin D (2000IU) orally once daily. Blood sample will be collected to measure serum vitamin D and calcium level at baseline. Then again blood sample will be collected to measure serum vitamin D level after 8 weeks of vitamin D administration. Regularity of medicine intake will be ensured over telephone, pill count, and from the patient's compliance sheet. The study has entails almost no potential risk to the patients. Patients would have every right to quit the experimental procedure any time during the experimentations if they desire each. However, it will be explained to them that the results of the present study may offer better prospects for similar patients in future, and that the present experimentations would carry no potential risk towards their health or their lives provided they strictly follow the instructions conducted to them.

ELIGIBILITY:
Inclusion Criteria:

* patients with MDD
* patients with PHQ - 9 score more than 10
* serum vitamin D less than 30 ng/ml
* Serum calcium level 8.5-10.5 mg/dl

Exclusion Criteria:

* Patients receiving antidepressant and dietary supplement with in last two months.
* Patients with other psychological disorder ( such as schizophrenia, bipolar affective disorder)
* Patients with parathyroid disease, thyroid disease, liver and kidney disease
* Patients with Diabetes mellitus

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2018-03-10 (Actual); Primary Completion 2019-01-10 (Estimated); Study Completion 2019-02-28 (Estimated)

PRIMARY OUTCOMES:
Severity of depression | 8 weeks
  Changes in severity of depression will be measured through the Patient Health Questionnaire - 9 (PHQ - 9) score at baseline and at 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- BSMMU, Dhaka, Bangladesh